CLINICAL TRIAL: NCT03818776
Title: A Pilot Trial of Proton Based Cardiac Sparing Accelerated Fractionated RadioTherapy in Unresectable Non-Small Cell Lung Cancer With Extended Durvalumab Therapy (PARTICLE-D)
Brief Title: Proton Based Cardiac Sparing Accelerated Fractionated RadioTherapy in Unresectable NSCLC
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Safety
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CASE1518
Record Dates: First submitted 2019-01-18; First posted 2019-01-28 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Durvalumab; PARTICLE-D
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab; Proton Therapy

STUDY DESIGN:
Intervention Model Description: Arm 1: 60 CGyE in 20 fractions (3+3 participants, 3-6 total) Arm 2: 69 CGyE in 23 fractions (3+3 participants, 3-6 total) Followed by expansion cohort at identified RP2 dose (12 participants)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Arm 1 - 60 CGyE in 20 fractions (Experimental): Proton based external beam radiation therapy with concurrent Durvalumab starting one week before RT.
  Radiation will follow dose escalation scheme:
  60 CGyE in 20 fractions (3+3 participants, 3-6 total)
  Interventions: Drug: Durvalumab; Radiation: Proton beam therapy RT
- Arm 2 - 69 CGyE in 23 fractions followed by expansion cohort a (Experimental): Proton based external beam radiation therapy with concurrent Durvalumab starting one week before RT.
  Radiation will follow dose escalation scheme:
  69 CGyE in 23 fractions (3+3 participants, 3-6 total) Followed by expansion cohort at identified RP2 dose (12 participants)
  Interventions: Drug: Durvalumab; Radiation: Proton beam therapy RT

INTERVENTIONS:
Drug: Durvalumab — Durvalumab (MEDI4736) is an anti-PD-L1 monoclonal antibody immunotherapy for lung cancer. Participants will receive 1500mg durvalumab via intravenous (IV) infusion Q4W for up to a maximum of 12 months (up to 13 doses/cycles) with the last administration on week 48 unless there is unacceptable toxicity, withdrawal of consent, or another discontinuation criterion is met. (N.b. If a participant's weight falls to 30kg (≤30 kg)), then the participant should receive weight-based dosing equivalent to 20 mg/kg of durvalumab Q4W after consultation between Investigator and Study Physician, until the weight improves to above 30 kg >30 kg, at which point the participant should start receiving the fixed dosing of durvalumab 1500 mg Q4W).
  Other Names: MEDI4736
Radiation: Proton beam therapy RT — Proton beam therapy is a type of RT where the proton stops at a specific depth according to its energy which allows for a sufficient tumor dose that may improve local control and survival while sparing normal organs at risk, such as the heart, lung, and spinal cord.

SUMMARY:
The purpose of this study is to treat participants with the combination of durvalumab (the study drug) and proton beam therapy. Proton beam therapy is a type of radiotherapy (RT) with a unique characteristic where the proton stops at a specific depth according to its energy. This may be advantageous in treating lung cancer because it allows for a sufficient tumor dose that may improve local control and survival while sparing normal organs at risk, such as the heart, lung, and spinal cord.

DETAILED DESCRIPTION:
All study participants will receive the same study intervention, which will consist of proton based external beam radiation therapy with concurrent Durvalumab starting one week before RT. Radiation will be delivered using cardiac sparing accelerated fractionated proton radiation. Radiation will have two dose escalation schemes followed by an expansion cohort for a total of approximately 24 participants enrolled at University Hospitals Cleveland Medical Center.

The objectives of this study are to evaluate the safety and feasibility of combination of durvalumab with two different schemes for accelerated fractionation proton radiation in participants who are unable to tolerate concurrent chemoradiation therapy. This will also include the evaluation of adverse events resulting from these treatment schemes.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status 0-2
* Body Weight >30kg
* Must have anticipated life expectancy of at least 12 weeks
* Must be histologically or cytologically confirmed to be non-small cell lung cancer (NSCLC) confirmed by biopsy within 90 days of registration.
* Any tumor PD-L1 expression is allowed (including 0% to 100%, or unknown at time of study enrollment)
* AJCC 8th Stage IIA-IIIC.
* Must be deemed by Specialist or tumor board decision to not be a candidate for surgical resection or the participant refuses resection. Being deemed unresectable can be for any reason, including but not limited to: tumor location, tumor characteristics, operative risks, poor participant lung function, participant age or medical comorbidity.
* Must be deemed by Medical Oncologist or tumor board decision to not be a candidate for or able to tolerate standard cisplatinum based doublet concurrent chemoradiation therapy or the participant refuses chemotherapy. Being deemed not a chemotherapy candidate can be for any reason, including but not limited to: age, medical comorbidity, end organ dysfunction.
* Pulmonary function testing performed within 365 days prior to registration. . Sufficient lung function as judged by the primary investigator based on anticipated radiation fields, with a minimum of FEV1 ≥ 0.7 Liter or ≥ 30% and DLCO ≥ 30% with or without bronchodilator within 365 days prior to registration.
* Adequate normal organ and marrow function as defined below:
* Haemoglobin ≥9.0 g/dL
* Absolute neutrophil count (ANC) 1.5 (or 1.0) x (> 1500 per mm3)
* Platelet count ≥75 x 109/L (>75,000 per mm3)
* Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). This will not apply to participants with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
* AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal
* Measured creatinine clearance (CL) >30 mL/min or Calculated creatinine CL>30 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:
* Males:

Creatinine CL (mL/min) = (Weight (kg) x (140 - Age)) / (72 x serum creatinine (mg/dL))

* Females:

Creatinine CL (mL/min) = (Weight (kg) x (140 - Age)) / (72 x serum creatinine (mg/dL)) x 0.85

* Subjects must have the ability to understand and the willingness to sign a written informed consent document.
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal participants. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:
* Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
* Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
* Participant is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

* Prior large field thoracic radiation therapy is not allowed except for at the discretion of the primary investigator. Prior SBRT to contralateral lung, or breast radiation greater than 3 years prior is allowed. Other prior thoracic radiation is allowed at the discretion of the primary investigator.
* Prior radiation therapy, or immunotherapy for current diagnosis of NSCLC
* Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
* Female participants who are pregnant or breastfeeding or male or female participants of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy.
* History of another primary malignancy except for:
* Malignancy treated with curative intent and with no known active disease ≥2 years before the first dose of IP and of low potential risk for recurrence
* Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
* Adequately treated carcinoma in situ (i.e. breast) without evidence of disease
* Low risk prostate cancer which has been treated or is undergoing active surveillance.
* Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria
* Participants with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
* Participants with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study Physician.
* Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP.
* Judgment by the investigator that the participant is unsuitable to participate in the study and the participant is unlikely to comply with study procedures, restrictions and requirements

Medication Specific Exclusion Criterion:

* History of primary immunodeficiency
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:
* Participants with vitiligo or alopecia
* Participants with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
* Any chronic skin condition that does not require systemic therapy
* Participants without active disease in the last 5 years may be included but only after consultation with the study physician
* Participants with celiac disease controlled by diet alone
* Participants with prior allogeneic bone marrow transplantation or prior solid organ transplantation
* Treatment with systemic immunosuppressive medications (including but not limited to prednisone > 10 mg daily, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [TNF] agents) within 2 weeks prior to Cycle 1, Day 1. However, the use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) for participants with orthostatic hypotension or adrenocortical insufficiency is allowed.
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the participant to give written informed consent
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis testing in line with local practice), hepatitis B (known positive hepatitis B surface antigen [HBsAg] result), hepatitis C, or human immunodeficiency virus (positive human immunodeficiency virus [HIV] 1/2 antibodies). Participants with a past or resolved hepatitis B (HBV) infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Participants positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Participants, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
* Prior randomisation or treatment in a previous durvalumab and/or tremelimumab clinical study regardless of treatment arm assignment.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-08-30 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-01-27 (Actual)

PRIMARY OUTCOMES:
Safety of intervention as defined by number of participants with Dose Limiting Toxicities (DLT) between first dose of Durvalumab and 30 days following completion of radiotherapy. | Up to 30 days following end of treatment
  Safety of intervention as defined by number of participants with DLT's between first dose of Durvalumab and 30 days following completion of radiotherapy. This is defined as 0 of 3 or 1 of 6 participants having no DLT of either Durvalumab or RT.
  DLT for RT defined as:
  1. Grade 4-5 non-hematologic serious adverse events (SAEs) considered by the Investigators to be probably or definitely related to protocol treatment.
  2. Grade 3 or higher cardiac adverse events (e.g. severely symptomatic congestive heart failure (CHF), myocarditis, pericardial effusion, myocardial infarction, symptomatic arrhythmia) considered by the Investigators to be probably or definitely related to protocol treatment.
  3. Grade 3 or higher pulmonary adverse events (e.g. dyspnea/pneumonitis) considered by the Investigators to be probably or definitely related to protocol treatment and not responsive to steroids.
  4. Failure to receive at least 54

SECONDARY OUTCOMES:
Feasibility of intervention defined by number of participants receiving full course of RT treatment and minimum of two doses of Durvalumab | Up to 30 days following end of treatment
  Feasibility of intervention is defined as a participant receiving the entire course of prescribed RT as well as having received a minimum of two doses of Durvalumab.
Number of participants with Adverse Events according to CTCAE v5.0 | Up to 30 days following end of treatment
  All toxicities will be graded according to NCI CTCAE, Version 5.0. See Adverse Events section.

CONTACTS AND LOCATIONS:
Overall Officials: Debora Bruno, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Will be shared with researchers who provide a methodologically sound proposal, to achieve aims in the approved proposal. To gain access, data requesters will need to sign a data access agreement